CLINICAL TRIAL: NCT03284125
Title: Lengthening Temporalis Myoplasty and Improvement of Primary Swallowing Disorders in Facial Paralysis
Acronym: MATPF
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/MATPF; 2017-A01577-46 (Other: IdRCB); 2017-39 (Other: CPP)
Record Dates: First submitted 2017-09-06; First posted 2017-09-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Peripheral Facial Paralysis
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Facial paralysis: Patients affected by facial paralysis treated by LTM The aim is to evaluate the improvement of the swallowing disorders after surgery.
  Interventions: Other: Swallowing disorders evaluation

INTERVENTIONS:
Other: Swallowing disorders evaluation — Self-administered questionnaires and non-invasive clinics tests

SUMMARY:
The facial paralysis is a frequent disease causing important functionals swallowing dysfunctions. The purpose of our study was to evaluate the improvement of the swallowing disorders after surgery by lengthening temporalis myoplasty (LTM) in the facial paralysis.

This prospective study has realised on the following of patients affected by facial paralysis treated by LTM. Self-administered questionnaires and clinics tests had realized to analyze three components oh the oral phase of the swallowing ( drooling, mastication and handicap). The evaluations was realized before the surgery and at 3 and 6 months after .

ELIGIBILITY:
Inclusion Criteria:

* Chronic peripheral facial paralysis
* Freyss score inferior at 15
* Benefiting of a lengthening temporalis myoplasty

Exclusion Criteria:

* Malformative syndrome
* Other swallowing trouble
* Psychiatric trouble
* Opposed at this study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients affected by facial paralysis and treated by lenthening temporalis myoplasty
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline lips pressure at 6 months | Baseline, 3 and 6 months
  Patients must contracted their lips of the paretic side in a manometer to evaluate the pressure of the lips before surgery and at 3 and 6 months after

SECONDARY OUTCOMES:
Drooling Severity and Frequency Scale (DSFS) | Baseline, 3 and 6 months
  The Drooling Score equals the sum of the Severity and Frequency sub-scores. the severity sub scores contains five items ( 1= never, 2= mild drooling, 3= moderate drool, 4= severe drool, 5= profuse drool) The frequency sub score contains four items ( 1= no drooling, 2= occasionally, 3=frequently, 4= constant drooling)
Visual scale of food residue | Baseline, 3 and 6 months
  Patients must eat a melba toast on paretic side and after we evaluate the food residue before surgery and at 3 and 6 months after
Dysphagia handicap index (DHI) | Baseline, 3 and 6 months
  This self-administered questionnaire allows to evaluate 3 types of handicap (physical, functional and social) It contains 30 questions and the maximum score is 120 (0= never, 1= almost never, 2= occasionally, 3= almost always, 4= always)

CONTACTS AND LOCATIONS:
Overall Officials: Boris LAURE, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Service de chirurgie maxillo-faciale, CHRU de TOURS, Tours, France

IPD SHARING:
Plan to Share IPD: No